CLINICAL TRIAL: NCT07166900
Title: Modified Thoracolumbar Interfascial Plane Block Versus Erector Spinae Plane Block For Enhancement Of Quality of Recovery After Lumbar Spine Surgery: A Prospective Randomized Controlled Study.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Ahmed sayed Shaban, Md, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: M800
Record Dates: First submitted 2025-09-09; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Espb (Active Comparator)
  Interventions: Procedure: Modified Thoracolumbar Interfascial Plane Block
- Tlib (Active Comparator)
  Interventions: Procedure: Modified Thoracolumbar Interfascial Plane Block

INTERVENTIONS:
Procedure: Modified Thoracolumbar Interfascial Plane Block — The TLIP block, introduced as a modification of the lumbar interfascial plane block, targets the dorsal rami of the thoracolumbar nerves by injecting local anesthetic into the fascial plane between the multifidus and longissimus muscles. This technique is designed to provide analgesia to the posterior elements of the spine, which are often the primary sources of pain after laminectomy

SUMMARY:
Aim of study The objective of the current study is to compare the efficacy of ultrasound-guided bilateral modified thoracolumbar interfascial plane (TLIP) block versus erector spinae (ES) block in optimizing early quality of recovery (QOR) following lumbar spine surgery under general anesthesia.

DETAILED DESCRIPTION:
Lumbar spine surgery, a common surgical procedure to alleviate spinal stenosis or disc herniation, is often associated with significant postoperative pain that can hinder early recovery and patient satisfaction. Effective pain management is critical to improve the quality of recovery (QOR), reducing complications, and facilitating early mobilization (1). Regional anesthesia techniques, such as nerve blocks, have gained popularity as part of multimodal analgesia strategies to minimize opioid use and enhance postoperative outcomes. Among these, the thoracolumbar interfascial plane (TLIP) block and the erector spinae (ES) block have emerged as promising ultrasound-guided techniques for managing pain after lumbar spine surgeries (2).

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for elective lumbar spine fixation 2-3 levels.
* American Society of Anesthesiologists(ASA) class I-III.

Exclusion Criteria:

* 1. Obese patients (Body Mass Index> 35). 2. Patients with neurological deficits, cardiopulmonary disease, hepatic or renal impairment.

  3. Patients with history of severe allergies to local anesthetics or other medications used during the procedure.

  4. Patients with history of coagulation disorder or anticoagulants. 5. Patients with emergency surgeries or re-do surgeries. 6. Patients with systemic infections or infections at the site of injection. 7. Patients with Psychiatric illnesses. 8. Patients with history of drug addiction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Quality of Recovery (QOR) | 24 hours postoperatively
  Assessed using the QOR-15 questionnaire at 24 hours postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Fayoum university hospital, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: No